CLINICAL TRIAL: NCT03865017
Title: A Safety and Tolerability Study of GB301 Given as a Single Intravenous Dose in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: A Safety and Tolerability Study of GB301
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VTBIO Co. LTD (Industry)
Collaborators: BHT Lifescience Austrailia Pty Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GB301-A01
Record Dates: First submitted 2019-02-15; First posted 2019-03-06 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-02

CONDITIONS: Alzheimer Disease
Keywords: Regulatory T cell; Treg; cell therapy; autologous
MeSH Terms: conditions — Alzheimer Disease | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regulatory T cells (Experimental): Biologicals: Autologous Regulatory T cells (1.7*10^5 cells/kg, i.v) other name: GB301
  Interventions: Biological: Regulatory T cells
- Placebo (Placebo Comparator): Saline+cell suspension solution infusion
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Regulatory T cells — The trial will be carried out in Alzheimer's disease patients. The investigators will isolate CD4+CD25+ Tregs from these patients, expand and injection.
  Other Names: GB301
  Arms: Regulatory T cells
Other: Saline — Saline+cell suspension solution infusion
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of multiple intravenous (IV) infusions at a single dose strength of GB301 in subjects with mild to moderate AD.

ELIGIBILITY:
Inclusion criteria:

1. Subjects who have voluntarily agreed to participate in the study and have signed a human research ethics committee-approved consent form after being briefed on the clinical study before undergoing any study-related procedure.
2. Male or female subjects aged ≥40 to ≤72 years with mild to moderate AD with an MMSE score at Screening and Baseline of ≥11.
3. Diagnostic confirmation by positron-emission tomography (PET) with florbetaben or another approved amyloid PET ligand. A previous amyloid imaging study with a positive result will be accepted. If none is available, then amyloid PET will be conducted during the Screening Period.
4. Subjects who have been clinically diagnosed with mild-to-moderate AD according to the 2011 version of the National Institute on Aging and Alzheimer's Association criteria and ≥6 month decline in cognitive function.
5. Subjects must have a caregiver/study partner who, in the opinion of the site principal investigator, has contact with the study subject for a sufficient amount of time (i.e. at least 6 hours per week) to provide informative responses on protocol assessments, and is willing and able to participate in all clinic visits. The legally acceptable representative (if appointed) and caregiver/study partner must provide written informed consent to participate in the study.
6. Formal education of ≥8 years.
7. Modified Hachinski Ischaemic Score ≤4 at Screening Visit.
8. The subject has had a documented computerized tomography or magnetic resonance imaging scan, interpreted by a radiologist or neurologist, within 36 months prior to randomization and after the subject met the National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association diagnostic criteria for probable AD. The scan must not show evidence for an alternative etiology for dementia.
9. No active depression and a Geriatric Depression Scale (15 items) score of ≤5.
10. Subjects should be generally healthy with mobility (ambulatory or ambulatory aided, i.e. walker or cane), vision and hearing (hearing aid permissible) sufficient for compliance with testing procedures.
11. Subject, if female, is postmenopausal (last natural menses ≥24 months) or has undergone a documented bilateral tubal ligation or hysterectomy. If last natural menses is <24 months, a serum follicle-stimulating hormone (FSH) value confirming post menopausal status should be employed, except if documentation of bilateral tubal ligation or hysterectomy is available.

    Women of childbearing potential need to apply at least 1 highly efficient contraceptive method.

    Male subject either agrees to use a highly efficient method of contraception if his female partner is of childbearing potential or must have been surgically sterilized prior to the Screening Visit.

    Highly efficient methods of contraception are defined as:
    * Hormonal methods such as oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full cycle before IP administration.
    * Total abstinence from sexual intercourse between the Screening Visit and 4 weeks after the last IP administration.
    * Intrauterine device.
    * Double barrier method (condoms, sponge, diaphragm, with spermicidal jellies, or cream).
12. Subjects with the capability of performing all cognitive and other tests required for this study in the opinion of the investigator.

Exclusion criteria:

1. Subjects who have taken drugs known to have or carry the potential for significant interactions with the IP within 14 days prior to the administration of this IP and during the study (e.g. non-specific immunosuppressive drugs, specific T cell immunosuppressive drugs, immunostimulants, immunomodulating agents) or any drugs that are considered unsuitable by investigator's judgment.
2. Subjects who have donated blood within 30 days prior to Screening or who have participated in clinical studies of other investigational medicinal products or commercially available drugs within 60 days prior to Screening.
3. Subjects who have experienced significant AEs or hypersensitivity to previous Treg therapy.
4. Subjects whom the investigator finds unsuitable for the clinical study participation based on clinically significant laboratory results, vital signs, ECG, or other examinations.
5. Subjects with a history of mental illness that may interfere with their participation in the clinical study, such as schizophrenia or bipolar affective disorder according to the investigator's judgment.
6. Subjects with any medical or neurological/neurodegenerative condition (other than AD) that, in the opinion of the investigator, might be a contributing cause to the subject's cognitive impairment or could lead to discontinuation, lack of compliance, interference with study assessments, or safety concerns.
7. Subjects who have had a stroke or transient ischemic attack or unexplained loss of consciousness in the past 1 year.
8. Subjects who have a history of clinically relevant brain hemorrhage, bleeding disorder, or cerebrovascular abnormalities.
9. Subjects with clinically relevant gastrointestinal, endocrine, inflammatory, or cardiovascular diseases that are not controlled by diet or medication.
10. Subjects with a history of alcohol or other substance abuse or dependence (with the exception of caffeine and nicotine) or a positive drug screen at Screening (amphetamines, barbiturates, cocaine, methamphetamine, methadone, opiates, phencyclidine, and tetrahydrocannabinol).
11. Subject has serum hepatitis, is a carrier of the hepatitis B virus surface antigen, is a carrier of the hepatitis C antibody, or is seropositive for human immunodeficiency virus antibodies as confirmed at Screening.
12. Subject has a history of cancer within 3 years of Screening with the exception of fully excised non-melanoma skin cancers or non-metastatic prostate cancer that has been stable for ≥6 months.
13. Subjects with uncontrolled hypertension with a resting systolic blood pressure exceeding 165 mmHg or diastolic blood pressure exceeding 96 mmHg.
14. Subjects with severe renal impairment (serum creatinine ≥1.7 mg/dL) at Screening.
15. Subjects with clinically relevant hepatic impairment (any of levels of alanine transaminase, aspartate transaminase, or bilirubin ≥2.0 times the upper limit of normal) at Screening.
16. Subjects who are taking or are expected to take a prohibited concomitant medication, such as steroid drugs and supplements that improve the blood circulation (e.g. omega-3 fatty acids) during the study. Concomitant medication affecting the central nervous system should be stable for ≥1 month before Screening and should not change during the study. Standard AD medication is permitted if initiated ≥3 months before enrollment and on a stable dose for ≥2 months.
17. Subjects who are unsuitable for participating in this clinical study for any other reason, based on the investigator's judgment.

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects With Clinically Significant Abnormalities in 12-lead Electrocardiogram | Between Baseline and 12 weeks
  The number of subjects with normal and abnormal ECG findings will be summarized for each treatment group at each time point. Clinical significance was determined by the investigator.
  ECG measures PR interval (ms), QRS interval, QT interval(ms), QTc interval (ms), and heart rate(bpm) for each treatment group at each time point.
Number of subjects with abnormal clinical chemistry parameters | Between Baseline and 12 weeks
  Blood samples will be collected for the assessment of following clinical chemistry parameters: Albumin, Total bilirubin, Total protein, Calcium, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN), Creatinine, Glucose, Sodium, Potassium, Chloride, Bicarbonate, LDH, FSH, Uricacid
Number of subjects with abnormal Hematology parameters | Between Baseline and 12 weeks
  Blood samples will be collected for the assessment of following hematology parameters: red blood cell (RBC) count, Hemoglobin, Hematocrit, mean corpuscular volume (MCV),mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), Platelet, white blood cell (WBC) count, Neutrophil, Lymphocyte, Monocyte, Eosinophil, Basophil
Number of subjects with abnormal Coagulation parameters | Between Baseline and 12 weeks
  Blood samples will be collected for the assessment of following coagulation parameters: Prothrombin Time(PT), International normalized ratio(INR), partial thromboplastin time (PTT)
Number of subjects with abnormal Urinalysis parameters | Between Baseline and 12 weeks
  Samples will be collected to measure specific gravity, potential of hydrogen (pH), glucose, protein, blood and ketones.
Number of subjects with abnormal vital signs | Between Baseline and 12 weeks
  Vital signs, including height (only assessed at Screening), weight, systolic and diastolic blood pressure, heart rate, and body temperature, will be measured after the subject has been in a sitting position for 5 minutes.
Number of subjects with abnormal vital signs | Between Baseline and 12 weeks
  Vital signs, including height (㎡, only assessed at Screening), weight(kg), systolic and diastolic blood pressure(mm Hg), heart rate(bpm), and body temperature(℃), will be measured after the subject has been in a sitting position for 5 minutes.
Number of subjects with adverse events (AEs) | Between Baseline and 12 weeks
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Number of subjects with abnormal physical examination | Between Baseline and 12 weeks
  A full physical examination will include assessments of the general apperance, skin, head, neck, eyes, ears, nose, throat, respiratory, cardiovascular, abdomen, extremities, musculoskeletal, neurological, lymph nodes etc.
Columbia Suicide Severity Rating Scale (C-SSRS) | Between Baseline and 12 weeks
  The C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. Some questions are yes/no and some are on a scale of 1 (low severity) to 5 (high severity). Completed suicide and non-fatal suicide events are yes/no questions and results presented are the number of participants with these events.

SECONDARY OUTCOMES:
Change from Baseline in Alzheimer´s Disease Assessment Scale- Cognitive Subscale (ADAS-Cog-13) Score | baseline, 29, 57, and 85 days
  13-item ADAS-Cog assesses a range of cognitive abilities including memory, comprehension, orientation in time and place, and spontaneous speech. Most items are evaluated by tests, but some are dependent on clinician ratings on a 5-point scale. The ADAS-Cog-13 is the ADAS-Cog-11 with 2 additional items: delayed word recall and total digit cancellation. Scores for the ADAS-Cog-13 range from 0 to 85 with higher scores indicating greater dysfunction.
Change from baseline in MMSE score | baseline, 29, 57, and 85 days
  The MMSE is a brief, screening instrument often used in clinical studies to assess dementia severity. The MMSE assesses several aspects of memory and cognitive functioning including orientation, attention, concentration, comprehension, recall, and praxis. The total possible score is 30, with high scores indicating less impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyoon Kim, Study Director — Director
Locations (1):
- Bht Lifescience Australia Pty Ltd, Brisbane, Queensland, Australia